CLINICAL TRIAL: NCT00415233
Title: Multicentre Randomised Trial of High Dose Versus Low Dose Radioiodine, With or Without Recombinant Human Thyroid Stimulating Hormone, for Remnant Ablation Following Surgery for Differentiated Thyroid Cancer [HILO]
Brief Title: High Dose vs Low Dose I 131 +/- rhTSH for Differentiated Thyroid Cancer
Acronym: HiLo
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UCL/05/83; CRUK-HILO-BRD/05/83 (Other Grant/Funding Number: Cancer Research UK); ISRCTN56078540 (Registry Identifier: ISRCTN); EU-20665; CTA-20363/0217/001/0001 (Other: Regulatory Authority Number); 2005-003687-37 (EudraCT Number)
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Cancer
Keywords: stage I follicular thyroid cancer; stage I papillary thyroid cancer; stage II follicular thyroid cancer; stage II papillary thyroid cancer; stage III follicular thyroid cancer; stage III papillary thyroid cancer; stage IV follicular thyroid cancer; stage IV papillary thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Thyrotropin; Thyrotropin Alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1.1Gbq with rhTSH (Experimental): Patients receive 1.1GBq dose of radioactive iodine and rhTSH
  Interventions: Biological: recombinant thyroid-stimulating hormone
- 3.2 GBq with rhTSH (Experimental): Patients receive 3.2GBq dose of radioactive idodine and rhTSH
  Interventions: Biological: recombinant thyroid-stimulating hormone
- 1.1GBq without rhTSH (Experimental): Patients only receive 1.1GBq dose of radioactive iodine and no rhTSH
  Interventions: Radiation: Radiodine ablation without rhTSH
- 3.2GBq without rhTSH (Experimental): Patients only receive 3.2GBq dose of radioactive iodine and no rhTSH
  Interventions: Radiation: Radiodine ablation without rhTSH

INTERVENTIONS:
Biological: recombinant thyroid-stimulating hormone — Recombinant thyroid stimulating hormone (rhTSH) should be given at a dose of 0.9mg by intramuscular injection on two consecutive days before ablation.
  Arms: 1.1Gbq with rhTSH; 3.2 GBq with rhTSH
Radiation: Radiodine ablation without rhTSH — Patients in this group do not receive rhTSH pre ablation.
  Arms: 1.1GBq without rhTSH; 3.2GBq without rhTSH

SUMMARY:
RATIONALE: Radioactive iodine uses radiation to kill tumor cells. Giving iodine I 131 with or without thyroid-stimulating hormone after surgery may kill any tumor cells that remain after surgery. It is not yet known which dose of iodine I 131 is more effective when given with or without thyroid-stimulating hormone in treating thyroid cancer.

PURPOSE: This randomized phase III trial is studying two different doses of iodine I 131 to compare how well they work when given with or without thyroid-stimulating hormone in treating patients who have undergone surgery for thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the percentage of successful remnant ablation at 6-8 months after administration of high- vs low-dose iodine I 131 with vs without recombinant thyroid-stimulating hormone in patients who have undergone total thyroidectomy for differentiated thyroid cancer.

Secondary

* Compare quality of life in patients treated with these regimens.
* Compare locoregional recurrence in patients treated with these regimens.
* Compare distant metastases, survival, and incidence of second primary malignancies in patients treated with these regimens.

OUTLINE: This is a multicenter, factorial, randomized study. Patients are stratified according to treatment center and disease stage (I vs II vs III vs IVA). Patients are randomized to 1 of 4 treatment arms.

Patients receive thyroid hormone replacement therapy (THRT)* with thyroxine (T4)** or liothyronine sodium (T3). Patients randomized to arm III or IV discontinue THRT 4 weeks (for patients receiving T4) or 2 weeks (for patients receiving T3) prior to remnant ablation.

NOTE: *Some treatment centers may chose to avoid starting THRT in patients randomized to arm III or IV.

NOTE: **Patients receiving T4 may be switched to T3 for 2 more weeks before discontinuing THRT.

* Arm I: Patients receive recombinant thyroid-stimulating hormone (rTSH) intramuscularly on days 1 and 2 and undergo remnant ablation with low-dose iodine I 131 on day 3.
* Arm II: Patients receive rTSH as in arm I and undergo remnant ablation with high-dose iodine I 131 on day 3.
* Arm III: Patients undergo remnant ablation with low-dose iodine I 131 as in arm I.
* Arm IV: Patients undergo remnant ablation with high-dose iodine I 131 as in arm II.

Quality of life is assessed at baseline, day 3 before remnant ablation, and at 3 months.

After completion of study therapy, patients are followed at 3 months, between 6-8 months, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 468 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed differentiated thyroid cancer

  * T1-T3, Nx, N0, N1, M0 disease
* Has undergone one- or two-stage total thyroidectomy with or without lymph node dissection

  * All known tumor resected (R0)
* Requires radioiodine remnant ablation

  * Does not require mandatory recombinant thyroid-stimulating hormone
* No Hurthle cell carcinoma or aggressive variants, including any of the following:

  * Tall cell, insular, poorly differentiated disease with diffuse sclerosing
  * Anaplastic or medullary carcinoma

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* No severe comorbid conditions including, but not limited to, any of the following:

  * Unstable angina
  * Recent heart attack or stroke
  * Severe labile hypertension
  * Dementia
  * Concurrent dialysis
  * Tracheostomy needing care
  * Learning difficulties
  * Inability to comply with radiation protection issues
  * Requirement for frequent nursing or medical supervision that puts staff at risk for unacceptable radiation exposure
* No other cancers except basal cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use effective contraception during and for 6 months after radioiodine remnant ablation
* Fertile male patients must use effective contraception during and for 4 months after radioiodine remnant ablation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 months since prior contrast CT scan
* No prior iodine I 131 or iodine I 123 pre-ablation scan
* No prior treatment for thyroid cancer (except surgery)

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with successful remnant ablation at 6-9 months | 6-9 months
  The percentage of patients who have a successful remnant ablation at 6-9 months after radioiodine administration.

SECONDARY OUTCOMES:
Quality of life as measured by the SF-36 questionnaire at baseline, the day of ablation, and at 3 months | Baseline to 3 months
  Quality of life as measured by the SF-36 questionnaire at baseline, the day of ablation, and at 3 months
Locoregional recurrence | During and post treatment
Distant metastases | Baseline to 5 years after randomisation of final patient
  After the 5 year follow up period, patients will be follwed at hospital according to routine practice.
Survival | Until patient death
Incidence of second primary malignancy | Baseline to 5 years after last patient is randomised
  After the 5 year follow up period, patients will be follwed at hospital according to routine practice.

CONTACTS AND LOCATIONS:
Overall Officials: Ujjal K. Mallick, MD, Study Chair — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (25):
- United Kingdom (25):
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Addenbrooke's Hospital, Cambridge, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Castle Hill Hospital, Cottingham, England
  - Derbyshire Royal Infirmary, Derby, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Ipswich Hospital, Ipswich, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Guy's Hospital, London, England
  - Royal Marsden - London, London, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - James Cook University Hospital, Middlesbrough, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Northampton General Hospital, Northampton, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Wales

REFERENCES:
- [Result] Mallick U, Harmer C, Yap B, Wadsley J, Clarke S, Moss L, Nicol A, Clark PM, Farnell K, McCready R, Smellie J, Franklyn JA, John R, Nutting CM, Newbold K, Lemon C, Gerrard G, Abdel-Hamid A, Hardman J, Macias E, Roques T, Whitaker S, Vijayan R, Alvarez P, Beare S, Forsyth S, Kadalayil L, Hackshaw A. Ablation with low-dose radioiodine and thyrotropin alfa in thyroid cancer. N Engl J Med. 2012 May 3;366(18):1674-85. doi: 10.1056/NEJMoa1109589. PMID 22551128
- [Derived] Dehbi HM, Mallick U, Wadsley J, Newbold K, Harmer C, Hackshaw A. Recurrence after low-dose radioiodine ablation and recombinant human thyroid-stimulating hormone for differentiated thyroid cancer (HiLo): long-term results of an open-label, non-inferiority randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Jan;7(1):44-51. doi: 10.1016/S2213-8587(18)30306-1. Epub 2018 Nov 27. PMID 30501974